CLINICAL TRIAL: NCT04636333
Title: Safety and Immunogenicity of a Recombinant COVID-19 Vaccine (CHO Cell) in Healthy Population Aged 18 Years and Older: A Phase I Study
Brief Title: Phase I Trial of a Recombinant COVID-19 Vaccine (CHO Cell)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Academy of Military Medical Sciences，Academy of Military Sciences，PLA (Unknown); ZHONGYIANKE Biotech Co, Ltd. (Unknown); LIAONINGMAOKANGYUAN Biotech Co, Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT096
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Safety; Tolerability; Immunogenicity; SARS-CoV-2 Vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Middle-dose vaccine (18-59 years) & Two dose regimen (Experimental): Two doses of middle-dose experimental vaccine at the schedule of day 0, 14.
  Interventions: Biological: Two doses of middle-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14
- Middle-dose vaccine (18-59 years) & Three dose regimen (Experimental): Three doses of middle-dose experimental vaccine at the schedule of day 0, 14 28.
  Interventions: Biological: Three doses of middle-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28
- High-dose vaccine (18-59 years) & Two dose regimen (Experimental): Two doses of high-dose experimental vaccine at the schedule of day 0, 14.
  Interventions: Biological: Two doses of high-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14
- High-dose vaccine (18-59 years) & Three dose regimen (Experimental): Two doses of High-dose vaccine at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28
- Middle-dose vaccine (> 59 years) & Three dose regimen (Experimental): Three doses of middle-dose experimental vaccine at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of middle-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28
- High-dose vaccine (> 59 years) & Three dose regimen (Experimental): Three doses of high-dose experimental vaccine at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28
- Middle-dose placebo (18-59 years) & Two dose regimen (Placebo Comparator): Two doses of middle-dose placebo at the schedule of day 0, 14.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 14 #middle-dose group#
- Middle-dose placebo (18-59 years) & Three dose regimen (Placebo Comparator): Three doses of middle-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28 #middle-dose group#
- High-dose placebo (18-59 years) & Two dose regimen (Placebo Comparator): Two doses of high-dose placebo at the schedule of day 0, 14.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 14 #High-dose group#
- High-dose placebo (18-59 years) & Three dose regimen (Placebo Comparator): Three doses of high-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28 #High-dose group#
- Middle-dose placebo (> 59 years) & Three dose regimen (Placebo Comparator): Three doses of high-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28 #middle-dose group#
- High-dose placebo (> 59 years) & Three dose regimen (Placebo Comparator): Three doses of high-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28 #High-dose group#

INTERVENTIONS:
Biological: Two doses of middle-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14 — Two doses of middle-dose (20µg/0.5ml) recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14.
  Arms: Middle-dose vaccine (18-59 years) & Two dose regimen
Biological: Three doses of middle-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28 — Three doses of middle-dose (20µg/0.5ml) recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28.
  Arms: Middle-dose vaccine (18-59 years) & Three dose regimen; Middle-dose vaccine (> 59 years) & Three dose regimen
Biological: Two doses of high-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14 — Two doses of high-dose (40µg/0.5ml) recombinant SARS-CoV-2 vaccine (CHOCell) at the schedule of day 0, 14.
  Arms: High-dose vaccine (18-59 years) & Two dose regimen
Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28 — Three doses of middle-dose (40µg/0.5ml) recombinant SARS-CoV-2 vaccine (CHO Cell) at the schedule of day 0, 14, 28.
  Arms: High-dose vaccine (18-59 years) & Three dose regimen; High-dose vaccine (> 59 years) & Three dose regimen
Biological: Two doses of placebo at the schedule of day 0, 14 #middle-dose group# — Two doses of placebo (0.5ml) at the schedule of day 0, 14.
  Arms: Middle-dose placebo (18-59 years) & Two dose regimen
Biological: Three doses of placebo at the schedule of day 0, 14, 28 #middle-dose group# — Three doses of placebo (0.5ml) at the schedule of day 0, 14, 28.
  Arms: Middle-dose placebo (18-59 years) & Three dose regimen; Middle-dose placebo (> 59 years) & Three dose regimen
Biological: Two doses of placebo at the schedule of day 0, 14 #High-dose group# — Two doses of placebo (0.5ml) at the schedule of day 0, 14.
  Arms: High-dose placebo (18-59 years) & Two dose regimen
Biological: Three doses of placebo at the schedule of day 0, 14, 28 #High-dose group# — Three doses of placebo (0.5ml) at the schedule of day 0, 14, 28.
  Arms: High-dose placebo (18-59 years) & Three dose regimen; High-dose placebo (> 59 years) & Three dose regimen

SUMMARY:
This is a phase I, randomized, placebo-controlled, double-blind study, to evaluate safety and immunogenicity of a recombinant SARS-CoV-2 vaccine (CHO cell) in Chinese healthy population aged 18 years and older. After randomization, the trial for each subject will last for approximately 13 months. Screening period is 1 week prior to randomization (Day -7 to Day -1), and each dose of either SARS-CoV-2 vaccine (CHO Cell) or placebo will be given intramuscularly (IM) on Day 0 and Day 14 for a two-dose regimen, or on Day 0, Day 14, and Day 28 for a three-dose regimen. Subjects who are ≥18 years old and ≤ 59 years old will be enrolled in adult group, and healthy elderly population who are >59 years old will be enrolled in elderly group. After adult group completes the follow-up 7 days after first vaccination, elderly group will be recruited.

DETAILED DESCRIPTION:
This is a phase I, randomized, placebo-controlled, double-blind study, to evaluate safety and immunogenicity of a recombinant SARS-CoV-2 vaccine (CHO cell) in Chinese healthy population aged 18 years and older. Healthy adults who are ≥18 years old and ≤59 years old will be enrolled in the adult group and healthy elderly population who are >59 years old will be enrolled in the elderly group. To ensure the enrollment of healthy subjects, screening tests (hematology, biochemistry, and urinalysis) will be performed prior to the vaccination. In the adults group, there are four regimen cohort: middle-dose at 0, 14 schedule, high-dose at 0, 14 schedule, middle-dose at 0,14, 28 schedule and high-dose at 0,14,28 schedule. In the elderly group, there are two regimen cohort: middle-dose at 0,14, 28 schedule and high-dose at 0,14,28 schedule. The subjects in regimen cohort will be randomized to receive vaccines or placebos at a ratio of 2:1.

The study will set up an Independent Data Monitoring Committee (IDMC) to conduct overall supervision. The IDMC is required to review the unblinded data when a significant event or risk occurs in the study that might cause the study to be suspended.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of ≥ 18 years old.
* The subject can understand and voluntarily sign the informed consent.
* The subject can The subject canprovide legal identification.

Exclusion Criteria:

* Have a history of close contact with a confirmed case of SARS-CoV-2, an asymptomatic infection in the previous 14 days, or a travel history/residential history in a community where a case has been reported.
* Have a history of contact with a person infected with SARS-CoV-2(a person with a positive nucleic acid test) in the previous 14 days.
* Patients with fever or respiratory symptoms who have been to middle or high-risk areas in the past 14 days or have exit history, or come from communities with case reports.
* In the past 14 days, there have been 2 or more cases of fever and/or respiratory symptoms in small areas such as homes, offices, school classes, etc.
* Have a history of SARS.
* Have a history of SARS-CoV-2 infection.
* Positive in SARS-CoV-2 IgG or IgM antibody screening.
* Positive in RT-PCR test of SARS-CoV-2 in throat swab.
* Positive in HIVantibody screening.
* Women who are breastfeeding, pregnant, or planning to become pregnant during the study period (based on the subject's self-report and blood pregnancy test results for women of childbearing age), or men who plan to conceive their partners during the study period.
* Subjects with body mass index (BMI) ≥35 kg/m2.
* Have a history of asthma, a history of vaccine or vaccine component allergy, have serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioedema.
* Subjects with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Subjects with autoimmune diseases or immunodeficiency/immunosuppression.
* Subjects with severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver and kidney diseases, malignant tumors, etc.
* Subjects with severe neurological disease (epilepsy, convulsions or convulsions) or mental illness.
* Subjects with thyroid disease or history of thyroidectomy, no spleen, functional asthenia, and any spleen or splenectomy caused by any condition.
* Abnormal blood coagulation function diagnosed by a doctor (such as coagulation factor deficiency, coagulopathy, abnormal platelet) or obvious bruise or coagulation disorder.
* Have received immunosuppressant therapy, cytotoxic therapy, and inhaled corticosteroids in the past 6 months (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis).
* Physical examination or chest CT imaging reveals clinically significant abnormalities.
* Abnormal laboratory test results such as hematology and biochemistry that are beyond the reference value range and have clinical significance.

  1. Routine blood test: white blood cell count, hemoglobin, platelet count.
  2. Blood biochemical index detection: alanine aminotransferase (ALT), aspartate aminotransferase (AST), fasting blood glucose, C-reactive protein, total bilirubin (TBIL), creatinine (CR), creatine phosphokinase (CPK).
  3. Urine routine indicators: urine protein (PRO), urine sugar, urine red blood cells.
  4. Coagulation function test: prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT), fibrinogen (FIB).
* Have a long history of alcohol or drug abuse.
* Received blood products within 3 months before receiving trial vaccine.
* Received other study drugs within 30 days before receiving the trail vaccine.
* Received a live attenuated vaccine within 14 days before receiving the experimental vaccine.
* Received a subunit or inactivated vaccine within 7 days before receiving the experimental vaccine.
* Various acute or chronic diseases occurred in the past 7 days.
* Axillary body temperature>37.0℃ before vaccination.
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

Exclusion criteria of subsequent dose:

If one of the following (1) to (4) adverse events (AE) occurs, the vaccination is prohibited, but other research steps can be continued according to the investigator's judgment; if one of the following (5), (6) adverse events occurs , The investigator will judge whether to inoculate; if one of the following events (7) to (10) occurs, the vaccination can be postponed within the time window specified in the plan.

* (1)The subjects used the same vaccine other than the experimental vaccine during the study.
* (2)Any serious adverse reactions that are causally related to vaccination.
* (3)Severe allergic or hypersensitivity reactions after vaccination (including urticaria/skin rash within 30 minutes after vaccination).
* (4)Any confirmed or suspected autoimmune disease or immunodeficiency disease, including human immunodeficiency virus (HIV) infection.
* (5)Acute or new-onset chronic disease after vaccination.
* (6)Other reactions (including severe pain, severe swelling, severe activity limitation, persistent high fever, severe headache, or other systemic or local reactions) are judged by the investigator.
* (7)Acute illness at the time of vaccination (Acute illness refers to moderate or severe illness with or without fever).
* (8)Axillary temperature >37.0℃ before vaccination.
* (9)Vaccination of subunit vaccine or inactivated vaccine within 7 days, live attenuated vaccine within 14 days.
* (10)According to the investigator's judgment, the subject has any other factors that are not suitable for vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-07-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of adverse reactions (AR) up to Day 28 after prime and boost vaccination of the recombinant SARS-CoV-2 vaccine (CHO cell) or placebo. | 28 days after first dose

SECONDARY OUTCOMES:
The proportion of adverse events (AE) within 7 days after each dose of the recombinant SARS-CoV-2 vaccine (CHO cell) or placebo. | 7 days after each dose
The proportion of abnormal markers of hematology, blood chemistry and urine analysis within 3 days after each dose of the recombinant SARS-CoV-2 vaccine (CHO cell) or placebo | 3 days after each dose
The proportion of serious adverse events up to Month 12 after prime and boost vaccination. | Month 12 after prime and boost vaccination
The proportion of neutralizing antibody positive conversion rate, positive rate, GMT and GMI at Day 14, Day 21, Day 28, Day 42 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo.#Day 0, Day 14 vaccination program# | Day 14, Day 21, Day 28, Day 42 after prime vaccination
The proportion of IgG antibody positive rate at Day 14, Day 21, Day 28, Day 42 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo.#Day 0, Day 14 vaccination program# | Day 14, Day 21, Day 28, Day 42 after prime vaccination
The proportion of neutralizing antibody positive conversion rate, positive rate, GMT and GM at Day 28, Day 35, Day 42, Day 56 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo.#Day 0, Day 14 ,Day 28 vaccination program# | Day 28, Day 35, Day 42, Day 56 after prime vaccination
The proportion of IgG antibody positive rate at Day 28, Day 35, Day 42, Day 56 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo.#Day 0, Day 14 ,Day 28 vaccination program# | Day 28, Day 35, Day 42, Day 56 after prime vaccination

OTHER OUTCOMES:
The proportion of IFN-γ secreted by T cells at Day 14 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo using ELISpot detection method | Day 14 after prime vaccination of recombinant SARS-CoV-2 vaccine (CHO cell) or placebo
Changes in serum cytokine (IL2, IL6) levels from baseline after 3 days of each dose | 3 days of each dose
  The units of IL2 and IL6 are both pg/ml
The proportion of neutralizing antibody and the GMT up to Month 3 after the whole process of vaccination | Month 3 after the whole process of vaccination
The proportion of neutralizing antibody and the GMT up to Month 6 after the whole process of vaccination | Month 6 after the whole process of vaccination
The proportion of neutralizing antibody and the GMT up to Month12 after the whole process of vaccination | Month 12 after the whole process of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Luo D, Pan H, He P, Yang X, Li T, Ning N, Fang X, Yu W, Wei M, Gao H, Wang X, Gu H, Mei M, Li X, Zhang L, Li D, Gao C, Gao J, Fei G, Li Y, Yang Y, Xu Y, Wei W, Sun Y, Zhu F, Hu Z, Wang H. A randomized, double-blind, placebo-controlled phase 1 and phase 2 clinical trial to evaluate efficacy and safety of a SARS-CoV-2 vaccine SCoK in adults. Clin Transl Med. 2022 Sep;12(9):e1016. doi: 10.1002/ctm2.1016. PMID 36103390